CLINICAL TRIAL: NCT04349943
Title: Effect of Standardized Nutritional Therapy on Clinical Prognosis and Cost-effectiveness of Inflammatory Bowel disease--a Prospective Study
Brief Title: Effect of Standardized Nutritional Therapy on Clinical Prognosis and Cost-effectiveness of Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YYK-2019001
Record Dates: First submitted 2019-12-25; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- inflammatory bowel disease (Experimental): According to the patient's disease condition, tube feeding time, internal and surgical diagnosis and treatment plan, standard step-based nutrition treatment was carried out for the patients with adaptive signs of nutrition treatment, and dynamic nutrition evaluation and efficacy evaluation were carried out.
  Interventions: Other: nutrition therapy

INTERVENTIONS:
Other: nutrition therapy — With enteral nutrition as the preferred solution, the gradual transition from slow to fast, from lean to dense, from essential to whole protein type is conducted.

SUMMARY:
To construct a standardized stepped nutritional treatment process for inpatients with inflammatory bowel disease, including nutritional risk screening and assessment, standardized nutritional treatment implementation, therapeutic effect follow-up and monitoring, family nutritional treatment follow-up, etc.

DETAILED DESCRIPTION:
Nutrition therapy of inflammatory bowel disease should follow the principle of sequential treatment of nutrition, which is the preferred scheme with enteral nutrition, from slow to fast, from weak to strong, from the elements to the whole protein on the steps of the gradual transition, in order to improve enteral nutrition in patients with tolerance and compliance and improve patient quality of life and long-term survival rate, reduce the social burden of disease, patients with good economic and social benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with inflammatory bowel disease

Exclusion Criteria:

* nothing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of nutritional status | 2 years
  We collect the body composition and grip strength of every IBD patients. Body composition include the muscle and fat contents.They are all measured as kilogram. (kg). Specific nutritional guidelines will be provided based on body composition results.
Improvement of quality of life | 2 years
  We asked each patient to complete the quality of life scale for every IBD patient. There are 32 questions in the scale, and each question has 7 options. The higher the score, the heavier it is.We will decide whether to give psychological intervention based on the score.

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hu'nan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-09-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04349943/Prot_000.pdf